CLINICAL TRIAL: NCT06029647
Title: Mangos to Reduce Cardiometabolic Risk Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California State Polytechnic University, Pomona (Other)
Responsible Party: Principal Investigator, Erik Froyen, PhD, Assistant Professor, California State Polytechnic University, Pomona
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 603036
Record Dates: First submitted 2023-08-26; First posted 2023-09-08 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2024-02

CONDITIONS: Healthy
MeSH Terms: interventions — Mangifera indica extract

STUDY DESIGN:
Intervention Model Description: The study will follow a randomized, controlled, crossover design with two 16-week dietary interventions separated by 4-week washout periods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mango (Experimental): The participants will consume one cup of fresh mango (100 kcal) per day for sixteen weeks.
  Interventions: Other: Mango
- Wafer (Placebo Comparator): The participants will consume vanilla wafers (100 kcal) per day for sixteen weeks.
  Interventions: Other: vanilla wafers

INTERVENTIONS:
Other: Mango — The participants will consume the treatment for 16 weeks, followed by a 4-week washout period.
  Arms: Mango
Other: vanilla wafers — vanilla wafers
  Arms: Wafer

SUMMARY:
This research study will determine the effects of mango consumption on blood pressure, body weight, dietary nutrient/pattern changes, total cholesterol, LDL-cholesterol, VLDL-cholesterol, triglycerides, and HDL-cholesterol in individuals with moderately elevated blood pressure and/or LDL-cholesterol.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of death in the United States and worldwide. Risk factors for CVD include, obesity, high serum concentrations of low-density lipoprotein (LDL) cholesterol, very-low-density lipoprotein (VLDL) cholesterol, triglycerides, and total cholesterol, as well as low serum concentrations of high-density lipoprotein (HDL) cholesterol. Hypertension (high blood pressure) is an additional risk factor for CVD. Dietary strategies to reduce the risk for CVD include consuming adequate amounts of fruits, vegetables, and whole grains. However, there is limited published research regarding the effects of specific food items on CVD risk factors. One such example are mangos; there are murine studies, but there is a paucity of human clinical trial research on the effects of mango consumption on decreasing the risk factors for CVD. Therefore, the objective of this proposed study will examine whether mango consumption lowers these CVD risk factors in individuals with hypertension and/or dyslipidemia. The hypothesis is that mango consumption will decrease LDL-cholesterol, VLDL-cholesterol, triglycerides, total cholesterol, body weight, and blood pressure, and increase HDL-cholesterol. This proposed study will follow a randomized, controlled, cross-over design. Blood draws will be performed at baseline, after 8 weeks, and at the end of each dietary treatment, at the Student Health Services at California State Polytechnic University, Pomona. In addition, height, body weight, and blood pressure measurements will be taken. Subsequently, lipid panels will be generated for each participant, and those with dyslipidemia and/or hypertension will consume either 1 cup of mango or vanilla wafers (iso-caloric control) per day for 16 weeks. After a 4-week washout period, the subjects will consume the other dietary treatment for 16 weeks. Two-way repeated measures Analysis of Variance (ANOVA), followed by least significant difference (LSD) post-hoc analysis, will be used to determine if there are significant differences in CVD risk factors between the mango and wafer diets. Furthermore, the participants will complete two 24-hour recalls during the week before each laboratory visit. It is expected that the consumption of mangos will decrease LDL-cholesterol, VLDL-cholesterol, triglycerides, total cholesterol, body weight, and blood pressure, and increase HDL-cholesterol compared to the wafer diet. This proposed study will be the first to determine the cardiovascular health benefits of mango consumption in humans.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy students (18 to 40 years)
* Attend California State Polytechnic University, Pomona
* Moderately elevated blood pressure (systolic greater than 120 mm Hg or diastolic greater than 80 mm Hg) and/or LDL-cholesterol (greater than 100 mg/dL)

Exclusion Criteria:

* Smokers
* Pregnancy
* Any medical issues
* Allergies or dislike of mangos
* Allergies to wheat, milk, eggs, and/or soy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2024-09-12 (Actual)

PRIMARY OUTCOMES:
Blood pressure (mm Hg) | 16 weeks for mango consumption and 16 weeks for vanilla wafer consumption
  Systolic and diastolic blood pressure will be measured.

SECONDARY OUTCOMES:
Body weight (kg) and height (cm) | 16 weeks for mango consumption and 16 weeks for vanilla wafer consumption
  Body weight, height, and body mass index (BMI) will be measured.
Blood lipids (mg/dL) | 16 weeks for mango consumption and 16 weeks for vanilla wafer consumption
  Total cholesterol, low-density lipoprotein cholesterol, very-low-density lipoprotein cholesterol, high-density lipoprotein cholesterol, and triglycerides will be measured.
Dietary analysis (six 24-hour dietary recalls per person in each treatment arm) | 16 weeks for mango consumption and 16 weeks for vanilla wafer consumption
  Dietary nutrient consumption will be measured (g or mg).

CONTACTS AND LOCATIONS:
Overall Officials: Erik Froyen, PhD, Principal Investigator — Cal Poly Pomona; Bonny Burns-Whitmore, DrPH, RD, Principal Investigator — Cal Poly Pomona
Locations (1):
- California State Polytechnic University, Pomona, Pomona, California, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share the data with other researchers.

REFERENCES:
- [Background] GBD 2017 Diet Collaborators. Health effects of dietary risks in 195 countries, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2019 May 11;393(10184):1958-1972. doi: 10.1016/S0140-6736(19)30041-8. Epub 2019 Apr 4. PMID 30954305
- [Background] Lee-Kwan SH, Moore LV, Blanck HM, Harris DM, Galuska D. Disparities in State-Specific Adult Fruit and Vegetable Consumption - United States, 2015. MMWR Morb Mortal Wkly Rep. 2017 Nov 17;66(45):1241-1247. doi: 10.15585/mmwr.mm6645a1. PMID 29145355
- [Background] Gorinstein S, Zemser M, Haruenkit R, Chuthakorn R, Grauer F, Martin-Belloso O, Trakhtenberg S. Comparative content of total polyphenols and dietary fiber in tropical fruits and persimmon. J Nutr Biochem. 1999 Jun;10(6):367-71. doi: 10.1016/s0955-2863(99)00017-0. PMID 15539312
- [Background] Papanikolaou Y, Fulgoni VL 3rd. Mango Consumption Is Associated with Improved Nutrient Intakes, Diet Quality, and Weight-Related Health Outcomes. Nutrients. 2021 Dec 24;14(1):59. doi: 10.3390/nu14010059. PMID 35010933
- [Background] Arshad F, Umbreen H, Aslam I, Hameed A, Aftab K, Al-Qahtani WH, Aslam N, Noreen R. Therapeutic Role of Mango Peels in Management of Dyslipidemia and Oxidative Stress in Obese Females. Biomed Res Int. 2021 Oct 23;2021:3094571. doi: 10.1155/2021/3094571. eCollection 2021. PMID 34725636
- [Background] Evans SF, Beebe M, Mahmood M, Janthachotikun S, Eldoumi H, Peterson S, Payton M, Perkins-Veazie P, Smith BJ, Lucas EA. Mango Supplementation Has No Effects on Inflammatory Mediators in Obese Adults. Nutr Metab Insights. 2017 Sep 25;10:1178638817731770. doi: 10.1177/1178638817731770. eCollection 2017. PMID 28983188
- [Background] O'Hara C, Ojo B, Emerson SR, Simenson AJ, Peterson S, Perkins-Veazie P, Payton ME, Hermann J, Smith BJ, Lucas EA. Acute Freeze-Dried Mango Consumption With a High-Fat Meal has Minimal Effects on Postprandial Metabolism, Inflammation and Antioxidant Enzymes. Nutr Metab Insights. 2019 Aug 19;12:1178638819869946. doi: 10.1177/1178638819869946. eCollection 2019. PMID 31452602
- [Background] Rosas M Jr, Pinneo S, O'Mealy C, Tsang M, Liu C, Kern M, Hooshmand S, Hong MY. Effects of fresh mango consumption on cardiometabolic risk factors in overweight and obese adults. Nutr Metab Cardiovasc Dis. 2022 Feb;32(2):494-503. doi: 10.1016/j.numecd.2021.11.001. Epub 2021 Nov 12. PMID 34953634
- [Background] Ross SM. African mango (IGOB131): a proprietary seed extract of Irvingia gabonensis is found to be effective in reducing body weight and improving metabolic parameters in overweight humans. Holist Nurs Pract. 2011 Jul-Aug;25(4):215-7. doi: 10.1097/HNP.0b013e318222735a. No abstract available. PMID 21697664